CLINICAL TRIAL: NCT00237575
Title: A Randomized Phase III Trial of Leukine® vs Neupogen® in Patients Receiving Cisplatin and Gemcitabine for Regionally Advanced or Metastatic Urothelial Cancer
Brief Title: Randomized Phase III Trial of Leukine® vs Neupogen® in Patients Receiving Cisplatin & Gemcitabine for Urothelial Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-GU-53B
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Bladder Cancer
Keywords: urothelial; bladder; gemcitabine; cisplatin; leukine; neupogen; filgrastim; sargramostim; metastatic; Regionally Advanced; Advanced
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Cisplatin; sargramostim; Filgrastim

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin
Drug: sargramostim
Drug: filgrastim

SUMMARY:
The main objective of this study is to compare the effectiveness of Leukine & Neupogen to decrease the incidence of grade 3 & 4 neutropenia in the treatment of patients receiving cisplatin & gemcitabine for urothelial (bladder) cancer.

All patients will receive chemotherapy with cisplatin plus gemcitabine in six 21-day cycles. Patients will also receive either Leukine (Arm A) or Neupogen (Arm B).

Patient Population: 100 patients will be enrolled (n=100) in this study. Patients cannot have undergone previous chemotherapy. Approximately 50 patients will be enrolled into each treatment arm.

Test Product, Dose, Mode of Administration: All patients will receive chemotherapy treatment with cisplatin (70 mg/kg) on Day 1 and gemcitabine (1000 mg/m2) on Days 1, 8, & 15 of each 21-day cycle. Patients will be randomized to receive either Leukine (250 µg/m2) or Neupogen (5 µg/kg) injected under the skin on Days 2-6, 9-13, & 16-20 of each cycle.

Duration of Treatment: Patients will receive a maximum of six 21-day cycles of treatment. The overall trial, including follow-up, is expected to be 3 years in duration.

DETAILED DESCRIPTION:
Objectives: To compare the efficacy of Leukine and Neupogen in the treatment of patients receiving cisplatin and gemcitabine for regionally advanced or metastatic urothelial cancer in regard to reduction of grade 3 and 4 neutropenia. Secondary objectives include a comparison of: hematologic and non-hematologic toxicities, anti-tumor effects, dose intensity, and quality of life in each treatment arm.

Methodology: The study will be a multi-institutional, randomized, phase III study in patients with regionally advanced or metastatic urothelial cancer. All patients will receive chemotherapy with cisplatin plus gemcitabine for six 21-day cycles. Patients will receive hematopoietic growth factor support with either Leukine (Arm A), or Neupogen (Arm B). Rates of anti-tumor responses and the incidence of toxicities in each treatment arm will provide a comparison of efficacy and safety for the hematopoietic support regimens.

Patient Population: Patients to be enrolled (n=100) in this study will have received a diagnosis of regionally advanced or metastatic urothelial cancer of the bladder, ureter, or renal pelvis and will have not undergone previous systemic chemotherapy. Approximately 50 patients will be enrolled into each treatment arm.

Main Criteria for Inclusion: Inclusion criteria for this study specify that patients have evaluable, biopsy-proven, surgically unresectable, regionally advanced, or metastatic urothelial cancer of the bladder, ureter, or renal pelvis. Additionally, patients must have an Eastern Cooperative Oncology Group performance status of 0-2 and adequate bone marrow, renal, and hepatic function. Patients who have undergone previous systemic chemotherapy will be excluded from this study.

Test Product, Dose, Mode of Administration: All patients will receive chemotherapeutic treatment with cisplatin (70 mg/kg) intravenously on Day 1 and gemcitabine (1000 mg/m2) intravenously on Days 1, 8, and 15 of each 21-day cycle. Patients will be randomized to receive either Leukine (250 µg/m2) or Neupogen (5 µg/kg) subcutaneously on Days 2-6, 9-13, and 16-20 of each cycle.

Duration of Treatment: Patients will receive a maximum of six 21-day cycles of treatment. The overall trial, including follow-up, is expected to be 3 years in duration.

Criteria for Evaluation: Efficacy will be assessed by, incidence of grade 3 and 4 toxicities, evaluation of complete and partial response, time to progression, overall and disease specific survival, planned vs administered doses, and quality of life. Safety will be assessed by, vital signs, physical examinations, clinical laboratory evaluations, and the reporting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, regionally advanced (T4b, N2, N3), or metastatic (M1) urothelial cancer of the bladder, ureter, or renal pelvis
* A minimum of one target lesion according to the RECIST criteria (Appendix D). Note: Bone metastases, leptomeningeal disease, ascites, pleural or pericardial effusions, lymphangitic spread or cystic lesions are not acceptable as target lesions.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Appendix B).
* Age >/=18 years or the age of majority in the state of the participating institution.
* Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter. Post menopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* An expected survival of at least four months.
* Adequate organ and marrow function as defined as follows:

  * leukocytes >/=3,000/µl,
  * absolute neutrophil count >/=1,500/µl,
  * hemoglobin >/=8.0g/dl,
  * platelets >/=100,000/µl,
  * total bilirubin and serum creatinine must be < 1.5 mg/dl
  * liver transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional ULN if alkaline phosphatase is </=ULN, or
  * alkaline phosphatase may be up to 4 x ULN if transaminases are </=ULN.
* Patients who have undergone previous radiation therapy or surgery may be enrolled into the study but such treatment must have been completed 4 or more weeks prior to entry to the study and the patient must have recovered. Further, patients who have undergone radiotherapy may not have received radiation to > 25% of the bone marrow. Previous intravesicular immunotherapy and chemotherapy are allowed.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Undergone previous systemic chemotherapy.
* Major surgery <4 weeks prior to study treatment start, or lack of complete recovery from major surgery.
* Participation in any investigational drug study within 4 weeks preceding treatment start.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be significant enough to preclude informed consent or interfering with compliance for oral drug intake.
* Previous history of cancer unless treatment was curative and completed >/=5 years prior to entry onto study, or unless diagnosed as one of the following: in situ carcinoma (any location), basal cell carcinoma, or non-metastatic squamous cell carcinoma of the skin.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled or untreated cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the teratogenic potential of cisplatin and gemcitabine. Lactating women are also excluded. (Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.)
* Peripheral neuropathy >/= grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of Leukine & Neupogen to prevent grade 3 & 4 neutropenia in patients receiving cisplatin & gemcitabine: assessed before cycles 3 & 5, then at end of treatment.
Safety of Leukine & Neupogen: evaluated before each cycle & blood work is evaluated weekly throughout the study.

SECONDARY OUTCOMES:
Reduction of grade 3 & 4 hematologic toxicities: evaluated weekly throughout the study.
Reduction of clinical hematologic toxicity including the # of: hospital days required for febrile neutropenia, transfusions & bleeding events, & days of outpatient antibiotics: evaluated throughout the study treatment and until resolved.
Reduction of non-hematologic toxicities: evaluated prior to each cycle.
Enhancement of anti-tumor effects (CR & PR, time to progression, OS & DFS): assessed before cycles 3 & 5, then on day 22 of cycle 6.
Dose intensity as planned vs administered: assessed during each treatment.
Quality of life: evaluated at baseline, pre-cylces 3 & 5, & end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Rinehart, MD, Study Chair — University of Kentucky
Locations (4):
- United States (4):
  - University of Louisville, Louisville, Kentucky
  - University of Nebraska, Omaha, Nebraska
  - New York Medical College, Hawthorne, New York
  - Montefiore Medical Center, The Bronx, New York